CLINICAL TRIAL: NCT01604902
Title: miRNAs and mRNAs in Psoriasis During Treatment With Biological Drugs.
Brief Title: miRNAs and mRNAs in Psoriasis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Aarhus (Other)
Collaborators: Abbott (Industry); Aage Bangs Fond (Other); Aase and Ejnar Danielsens Foundation (Other); Direktør Jacob Madsens Og Hustru Olga Madsens Fond (Unknown); Snedkermester Sophus Jacobsen and hustru Astrid Jacobsens Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: 2011-218/2-86
Record Dates: First submitted 2012-05-22; First posted 2012-05-24 (Estimated); Last update posted 2014-08-25 (Estimated); Status verified 2013-01

CONDITIONS: Psoriasis
Keywords: Psoriasis mRNA and miRNA
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — tissue: 4mm skin pinch biopsies for mRNA and miRNA extration.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Psoriasis vulgaris: Patients with psoriasis vulgaris who are going to be treated with biological drugs independent of this project(according to national guidelines).
  Interventions: Other: 4 mm punch biopsies

INTERVENTIONS:
Other: 4 mm punch biopsies — 4 mm punch-biopsies from lesional and non-lesional psoriatic skin at day 0 and up to four times after treatment at the following days: 4, 14, 28 or 84.

SUMMARY:
PURPOSE - The purpose of this study is to identify and determine miRNA expression and their targets before and during biological treatment of psoriatic patients.

HYPOTHESIS - Changes in the expression of specific miRNAs play an important role for the cytokine expression profile seen in lesional psoriatic skin. miRNAs may therefore serve as a potential target for future anti-psoriatic treatment as well as possible predictors of biological treatment response.

PERSPECTIVES - The results from this novel research project will increase the investigators understanding of the underlying mechanisms leading to psoriasis. Furthermore it is possible that predictors of treatment response can be identified. Identification of biomarkers predicting treatment outcome will individualize patient care, reduce number of treatment failures and thereby have a tremendous socio-economic impact and increase the patients quality of life.

DETAILED DESCRIPTION:
BACKGROUND: Psoriasis is a chronic inflammatory skin disease affecting 2-3% of the population worldwide and having tremendously impact on the patients' quality of life. Progress has been made in the understanding of the cellular immunology and biology of psoriasis, but the ultimate cause for psoriasis is still unknown.

miRNA are ~22 nt noncoding RNAs that modulate gene expression at the post-transcriptional level. miRNAs have regulatory roles in development, differentiation, growth control and apoptosis.

AIM OF PROJECT: To identify psoriasis specific miRNA. To investigate the differences in miRNA expression and their targets between lesional and non-lesional psoriatic skin. To investigate changes in the miRNA expression during biological treatment.

METHODS: Patients included are adults (> 18 years) with psoriasis vulgaris who are going to be treated with biological drugs independent of this project (according to national guidelines). A signed informed consent will be obtained before patients are included in the project.

Patients are not allowed to have received local treatment 2 weeks before inclusion or having had any systemic treatment including UVB 6 weeks before inclusion. 4 mm punch-biopsies from lesional and non-lesional psoriatic skin will be obtained using a local anaesthetic containing 1% Lidocaine at day 0 and up to four times after treatment at the following days 4, 14, 28 or 84. Before and during treatment patients will be monitored with a clinical score including PASI, BSA and PGA. Clinical evaluation will be conducted by a trained dermatologist at day 0 and day 84. That allows us to compare clinical changes to findings obtained during this study.

miRNA and mRNA expression will be analysis with quantitativePCR, protein level with ELISA and cell proliferation will be measure by a standard cell proliferation assay. miRNA microarray are commercially available and will be used to identify miRNA of interest.

NOVELTY: Changes in the expression of miRNA in psoriasis and miRNA regulation during treatment of psoriasis have only been sparsely studied. The results from this research project will therefore increase our understanding of the underlying mechanisms leading to psoriasis and may generate important new tools for individualised treatment of psoriasis.

ELIGIBILITY:
Inclusion Criteria:

* Males and females aged 18 or above
* Patients with psoriasis vulgaris who are going to be treated with biological drugs independent of this project.
* A signed informed consent form prior of any study-mandated procedure.

Exclusion Criteria:

* No local treatment 2 weeks before inclusion
* No systemic treatment including UVB 6 weeks before inclusion.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients included are adults (> 18 years) with psoriasis vulgaris who are going to be treated with biological drugs independent of this project.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2011-03; Primary Completion 2015-03 (Estimated); Study Completion 2016-01 (Estimated)

PRIMARY OUTCOMES:
miRNA and mRNA regulation in psoriatic skin | jan 2015

CONTACTS AND LOCATIONS:
Overall Officials: Line R OIsen, MD, Principal Investigator — Aarhus University Hospital
Locations (1):
- Aarhus University Hospital, Aarhus, Region Midt, Denmark